CLINICAL TRIAL: NCT03394287
Title: A Phase II, Open-labeled, Randomised, Non-comparative, Two-arms Investigator-initiated Clinical Trial of SHR-1210 (Anti-PD-1 Antibody) in Combination With Apatinib in Subjects With Advanced Triple Negative Breast Cancer
Brief Title: A Trial of SHR-1210 (an Anti-PD-1 Antibody) in Combination With Apatinib in Patients With Advanced TNBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Erwei Song, M.D., Ph.D., President of Sun Yat-sen Memorial Hospital, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-APTN-IIT-TNBC
Record Dates: First submitted 2018-01-02; First posted 2018-01-09 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210 +Apatinib daily dosing (Experimental): SHR-1210 200mg(3mg/kg for patient whose weight is below 50kg) iv Q2W combination With Apatinib 250mg, po, daily dosing (d1-d14)
  Interventions: Drug: SHR-1210; Drug: Apatinib
- SHR-1210+Apatinib intermittent dosing (Experimental): SHR-1210 200mg (3mg/kg for patient whose weight is below 50kg) iv Q2W combination With Apatinib 250mg, po, intermittent dosing(Continuous administration for 7 days every 14 days, d1-d7)
  Interventions: Drug: SHR-1210; Drug: Apatinib

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 200mg (3mg/kg for patient whose weight is below 50kg) will be administered as an intravenous infusion over 30 minutes every two weeks until unacceptable toxic effects or disease progression or other termination criteria appeared.
Drug: Apatinib — Apatinib 250mg will be taked daily/intermittent dosing until unacceptable toxic effects or disease progression or other termination criteria appeared.

SUMMARY:
This is a Phase II, Open-labeled, Randomised, Parallel, Non-comparative, Two-arms, Investigator-initiated Clinical Trial of SHR-1210 (Anti-PD-1 Antibody) in Combination With Apatinib (VEGFR2 inhibitor) in Subjects with Advanced Triple Negative Breast Cancer. Subjects with advanced Triple Negative Breast Cancer will be recruited. Patients will be randomised to two treatment arms of this study. One arm is SHR-1210 combination with apatinib daily dosing, and the other arm is SHR-1210 combination with apatinib intermittent dosing; each arm will enrolle10-29 subjects (Simons two stage design).

This study aims to evaluate the efficacy and safety of SHR-1210 combination with apatinib in the treatment of advanced TNBC.

ELIGIBILITY:
Inclusion Criteria:

* The patients signed the written informed consent
* Women aged 18-70.
* The pathologic diagnosis of recurrent metastatic triple negative breast cancer ［ER-negative(IHC<1%), PR-negative(IHC<1%), HER2-negative（IHC-/+ or IHC++ and FISH/CISH-）］.
* At least one measuring lesion that conforms to RECIST v1.1 standard.
* The number of chemotherapy lines in the metastatic phase was <3 line.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
* Have a life expectancy of at least 12 weeks.
* Female Subjects of childbearing potential must have a negative serum pregnancy test within 72 hours before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 3 months after the last dose of study treatment.
* The patients can swallow pills.
* The results of patients' blood tests are as follows: • Hb≥90g/L; • Plt≥90E+9/L; • Neutrophils≥1.5E+9/L; • ALT and AST ≤ triple of normal upper limit; • TBIL ≤ 1.5 times of normal upper limit; • Creatinine ≤ 1.5 times of normal upper limit.

Exclusion Criteria:

* The subjects had any history of autoimmune disease or any use of systemic glucocorticoid or immunosuppressive medications.
* Subjects with severe allergic reactions to other monoclonal antibodies.
* The subjects had a central nervous system metastases with clinical symptoms.
* History of hypertension and antihypertensive medications are not well controlled.
* A heart condition or disease that is not well controlled.
* Subjects had active infections or recent treatment with a systemic immunostimulatory agent (received within the previous 4 weeks).
* Other clinical trials of drugs were used in the first four weeks of the first medication.
* Subjects with treatment history of anti-angiogenesis drugs or check-point inhibitors.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
ORR | from the first drug administration up to the first occurrence of progression or death(up to 24 months)
  Overall Response Rate

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | from the first drug administration to within 90 days for the last SHR-1210 dose
  adverse events/serious adverse events
DCR | from the first drug administration up to the first occurrence of progression or death(up to 24 months)
  Disease Control Rate
DoR | from the first drug administration up to the first occurrence of progression or death(up to 24 months)
  Duration of response
PFS | from the first drug administration up to the first occurrence of progression or death (up to about 5 years)
  Progression-Free-Survival
One year-OS | 12 months after the first drug administration
  One year-Overall survival
CBR | from the first drug administration up to the first occurrence of progression or death(up to 24 months)
  Clinical benefit rate
TTR | from the first drug administration up to one year
  Time to response
Frequencies Of Biomarkers | pre-dose, and up to two years
  Biomarkers (PD-L1, PD-1, VEGF-A, eg) in tumor tissue and peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu J, Liu Q, Li Y, Li Q, Su F, Yao H, Su S, Wang Q, Jin L, Wang Y, Lau WY, Jiang Z, Song E. Efficacy and safety of camrelizumab combined with apatinib in advanced triple-negative breast cancer: an open-label phase II trial. J Immunother Cancer. 2020 May;8(1):e000696. doi: 10.1136/jitc-2020-000696. PMID 32448804